CLINICAL TRIAL: NCT01725269
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Intermediate/Long Term Safety and Efficacy of AIR001 in Subjects With WHO Group 1 Pulmonary Arterial Hypertension
Brief Title: Long-term Study of AIR001 in Subjects With WHO Group 1 Pulmonary Arterial Hypertension Who Completed AIR001-CS05
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early dt acquisition of Sponsor and change in corporate priorities
Sponsor: Aires Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIR001-CS06
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: AIR001; sodium nitrite; PAH; Pulmonary Arterial Hypertension; inhaled sodium nitrite
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 80mg AIR001, nebulized four times daily (Experimental): AIR001, 80 mg into nebulizer
  Interventions: Drug: AIR001
- 46 mg AIR001, nebulized four times daily (Experimental): AIR001, 46 mg into nebulizer
  Interventions: Drug: AIR001
- 80mg AIR001, nebulized once daily (Experimental): AIR001, 80 mg into nebulizer
  Interventions: Drug: AIR001

INTERVENTIONS:
Drug: AIR001 — All doses specified are the amount loaded into the I-neb AAD System nebulizer.
  Other Names: (sodium nitrite inhalation soution)

SUMMARY:
The AIR001-CS05 study evaluated the safety and efficacy (effectiveness) of AIR001 over 16 weeks in subjects who have PAH. The purpose of the AIR001-CS06 study is to evaluate the intermediate / long-term safety of AIR001 in subjects who have completed the AIR001-CS05 study. Assessments to evaluate the effectiveness of the study drug will include measurements of exercise ability and evaluations of PAH disease symptoms.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the intermediate/long-term safety of inhaled nebulized AIR001 administered according to 3 treatment arms (80 milligrams (mg) 4 times daily, 46 mg 4 times daily, or 80 mg once daily) in subjects with World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH) who have completed the 16-week AIR001-CS05 study.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study prior to initiation of any subject-mandated procedures.
2. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Has completed the 16-week AIR001-CS05study as planned.
4. If on corticosteroids, has been receiving a stable dose of less than or equal to 20 mg/day of prednisone (or equivalent dose, if other corticosteroid) for at least 1 month (30 days) prior to the AIR001-CS05 study Baseline/Day 1 visit. If receiving treatment for Connective Tissue Disease (CTD) with any other drugs, doses should remain stable, if clinically feasible, for the duration of the AIR001-CS06 study.
5. Women of childbearing potential must be using at least one form of medically acceptable contraception (i.e. either oral, topical, implanted hormonal contraceptives, or an intrauterine device) or two barrier methods; have a negative pregnancy test at Screening and Baseline/Day 1 and agree to use reliable methods of contraception until at least 24-hours after the last dose of study drug. Women who are surgically sterile (i.e. hysterectomy, bilateral oophorectomy, or tubal ligation) or those who are post-menopausal for at least 2 years are not considered to be of childbearing potential. Men who are not sterile (i.e. have not had a vasectomy) must also agree to use contraception until at least 24-hours after the last dose of study drug.

Exclusion Criteria:

1. Participation in a device or other interventional clinical studies (other than AIR001-CS05), within 1 month (30 days) of Baseline/Day 1 and/or during study participation.
2. Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure > 160 mmHg or sitting diastolic blood pressure > 100 mmHg during Baseline/Day 1 visit.
3. Systolic blood pressure < 90 mmHg at Baseline/Day 1.
4. Diagnosis of Down syndrome.
5. Moderate to severe hepatic impairment classified as a Child-Pugh Class B or C at Baseline/Day 1.
6. Has chronic renal insufficiency as defined by serum creatinine > 2.5 mg/dL or has an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min at Baseline/Day 1, or requires dialytic support.
7. Has a hemoglobin (Hgb) concentration < 8.5 g/dL at Baseline/Day 1.
8. Personal or family history of the following:

   1. Congenital or acquired methemoglobinemia;
   2. RBC CYPB5 reductase deficiency.
9. History of glucose-6-phosphate dehydrogenase (G6PD) deficiency or any contraindication to receiving methylene blue.
10. For subjects with Human immunodeficiency virus (HIV) associated PAH, requirement for the use of inhaled pentamidine.
11. The use of oral or topical nitrates (nitroglycerin, glyceryl trinitrate (GTN), isosorbide dinitrate, and isosorbide mononitrate) within 1 month (30 days) prior to Baseline/Day 1 or throughout the AIR001-CS06 study until EOS or Termination visit. Note: Intravenous GTN in an emergency setting may be administered by starting with a low dose and titrating upward, while the subject is being monitored closely for changes in blood pressure and heart rate.
12. Known or suspected hypersensitivity or allergic reaction to sodium nitrite or sodium nitrate.
13. History of malignancy within 5-years prior to Baseline/Day 1 of the AIR001-CS05 study, with the exception of localized non-metastatic basal cell carcinoma of the skin and in situ carcinoma of the cervix.
14. Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
15. Has a psychiatric, addictive or other disorder that compromises the ability to give informed consent for participating in this study. This includes subjects with a recent history of abusing alcohol or illicit drugs 1 month (30 days) prior to study Baseline/Day 1 of the AIR001-CS05 study and for the duration of the study.
16. Is currently pregnant or breastfeeding or intends to become pregnant during the duration of the study.
17. Investigators, study staff or their immediate families.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the intermediate/long-term safety of inhaled nebulized AIR001 | minimum of 6 months
  The primary objective of this study is to evaluate the intermediate/long-term safety of inhaled nebulized AIR001 administered according to 3 treatment arms (80 milligrams (mg) 4 times daily, 46 mg 4 times daily, or 80 mg once daily) in subjects with World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH) who have completed the 16-week AIR001-CS05 study.

SECONDARY OUTCOMES:
To assess the effect of inhaled AIR001 on Time to Clinical Worsening, 6MWD, Functional Class, and Quality of Life | minimum of 6 months
  The secondary objectives of this study are to evaluate the effect of inhaled nebulized AIR001 administered according to 3 different treatment arms (80 mg 4 times daily, 46 mg 4 times daily, or 80 mg once daily) in subjects with WHO Group 1 PAH who completed the 16-week AIR001-CS05 study, as determined by time to the first morbidity/mortality event as defined in Time to Clinical Worsening (TTCW) assessments and by change from Baseline in AIR001-CS05 to the 40th week from the start of AIR001 nebulization in AIR001-CS05 (Week 24 of AIR001-CS06) and End of Study (EOS) or Termination visit of AIR001-CS06 in the following:6-Minute Walk Distance (6MWD) assessed at peak, WHO/NYHA Functional Class, Quality of Life (QOL) as measured by SF-36,Borg Dyspnea Index,6MWD assessed at trough

CONTACTS AND LOCATIONS:
Overall Officials: Adaani E Frost, M.D., Principal Investigator — Baylor College of Medicine, Houston
Locations (25):
- United States (17):
  - UCSD Medical Center, La Jolla, California
  - UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Adaani Frost, M.D., Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (4):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
- Hungary (4):
  - Gottsegen Gyorgy Hungarian, Budapest
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
  - University of Szeged, Szeged

REFERENCES:
- [Background] Ahanchi SS, Tsihlis ND, Kibbe MR. The role of nitric oxide in the pathophysiology of intimal hyperplasia. J Vasc Surg. 2007 Jun;45 Suppl A:A64-73. doi: 10.1016/j.jvs.2007.02.027. PMID 17544026
- [Background] Zuckerbraun BS, George P, Gladwin MT. Nitrite in pulmonary arterial hypertension: therapeutic avenues in the setting of dysregulated arginine/nitric oxide synthase signalling. Cardiovasc Res. 2011 Feb 15;89(3):542-52. doi: 10.1093/cvr/cvq370. Epub 2010 Dec 22. PMID 21177703
- [Background] Williamson DJ, Wallman LL, Jones R, Keogh AM, Scroope F, Penny R, Weber C, Macdonald PS. Hemodynamic effects of Bosentan, an endothelin receptor antagonist, in patients with pulmonary hypertension. Circulation. 2000 Jul 25;102(4):411-8. doi: 10.1161/01.cir.102.4.411. PMID 10908213
- [Background] Alef MJ, Vallabhaneni R, Carchman E, Morris SM Jr, Shiva S, Wang Y, Kelley EE, Tarpey MM, Gladwin MT, Tzeng E, Zuckerbraun BS. Nitrite-generated NO circumvents dysregulated arginine/NOS signaling to protect against intimal hyperplasia in Sprague-Dawley rats. J Clin Invest. 2011 Apr;121(4):1646-56. doi: 10.1172/JCI44079. Epub 2011 Mar 23. PMID 21436585
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Badesch DB, Champion HC, Gomez Sanchez MA, Hoeper MM, Loyd JE, Manes A, McGoon M, Naeije R, Olschewski H, Oudiz RJ, Torbicki A. Diagnosis and assessment of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S55-S66. doi: 10.1016/j.jacc.2009.04.011. PMID 19555859
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Barbosa PB, Ferreira EM, Arakaki JS, Takara LS, Moura J, Nascimento RB, Nery LE, Neder JA. Kinetics of skeletal muscle O2 delivery and utilization at the onset of heavy-intensity exercise in pulmonary arterial hypertension. Eur J Appl Physiol. 2011 Aug;111(8):1851-61. doi: 10.1007/s00421-010-1799-6. Epub 2011 Jan 12. PMID 21225278
- [Background] Battistini B, Berthiaume N, Kelland NF, Webb DJ, Kohan DE. Profile of past and current clinical trials involving endothelin receptor antagonists: the novel "-sentan" class of drug. Exp Biol Med (Maywood). 2006 Jun;231(6):653-95. PMID 16740981
- [Background] Battle RW, Davitt MA, Cooper SM, Buckley LM, Leib ES, Beglin PA, Tischler MD. Prevalence of pulmonary hypertension in limited and diffuse scleroderma. Chest. 1996 Dec;110(6):1515-9. doi: 10.1378/chest.110.6.1515. PMID 8989070
- [Background] Chaouat A, Bugnet AS, Kadaoui N, Schott R, Enache I, Ducolone A, Ehrhart M, Kessler R, Weitzenblum E. Severe pulmonary hypertension and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 15;172(2):189-94. doi: 10.1164/rccm.200401-006OC. Epub 2005 Apr 14. PMID 15831842
- [Background] Clozel M, Breu V, Gray GA, Kalina B, Loffler BM, Burri K, Cassal JM, Hirth G, Muller M, Neidhart W, et al. Pharmacological characterization of bosentan, a new potent orally active nonpeptide endothelin receptor antagonist. J Pharmacol Exp Ther. 1994 Jul;270(1):228-35. PMID 8035319
- [Background] Farber HW, Loscalzo J. Pulmonary arterial hypertension. N Engl J Med. 2004 Oct 14;351(16):1655-65. doi: 10.1056/NEJMra035488. No abstract available. PMID 15483284
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Background] Ghofrani HA, Barst RJ, Benza RL, Champion HC, Fagan KA, Grimminger F, Humbert M, Simonneau G, Stewart DJ, Ventura C, Rubin LJ. Future perspectives for the treatment of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S108-S117. doi: 10.1016/j.jacc.2009.04.014. PMID 19555854
- [Background] Giaid A, Saleh D. Reduced expression of endothelial nitric oxide synthase in the lungs of patients with pulmonary hypertension. N Engl J Med. 1995 Jul 27;333(4):214-21. doi: 10.1056/NEJM199507273330403. PMID 7540722
- [Background] Gielis JF, Lin JY, Wingler K, Van Schil PE, Schmidt HH, Moens AL. Pathogenetic role of eNOS uncoupling in cardiopulmonary disorders. Free Radic Biol Med. 2011 Apr 1;50(7):765-76. doi: 10.1016/j.freeradbiomed.2010.12.018. Epub 2010 Dec 21. PMID 21172428
- [Background] Gladwin MT, Raat NJ, Shiva S, Dezfulian C, Hogg N, Kim-Shapiro DB, Patel RP. Nitrite as a vascular endocrine nitric oxide reservoir that contributes to hypoxic signaling, cytoprotection, and vasodilation. Am J Physiol Heart Circ Physiol. 2006 Nov;291(5):H2026-35. doi: 10.1152/ajpheart.00407.2006. Epub 2006 Jun 23. PMID 16798825
- [Background] Gladwin MT, Vichinsky E. Pulmonary complications of sickle cell disease. N Engl J Med. 2008 Nov 20;359(21):2254-65. doi: 10.1056/NEJMra0804411. No abstract available. PMID 19020327
- [Background] Hassoun PM, Mouthon L, Barbera JA, Eddahibi S, Flores SC, Grimminger F, Jones PL, Maitland ML, Michelakis ED, Morrell NW, Newman JH, Rabinovitch M, Schermuly R, Stenmark KR, Voelkel NF, Yuan JX, Humbert M. Inflammation, growth factors, and pulmonary vascular remodeling. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S10-S19. doi: 10.1016/j.jacc.2009.04.006. PMID 19555853
- [Background] Humbert M, Morrell NW, Archer SL, Stenmark KR, MacLean MR, Lang IM, Christman BW, Weir EK, Eickelberg O, Voelkel NF, Rabinovitch M. Cellular and molecular pathobiology of pulmonary arterial hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):13S-24S. doi: 10.1016/j.jacc.2004.02.029. PMID 15194174
- [Background] Humbert M, Sitbon O, Simonneau G. Treatment of pulmonary arterial hypertension. N Engl J Med. 2004 Sep 30;351(14):1425-36. doi: 10.1056/NEJMra040291. No abstract available. PMID 15459304
- [Background] Hunter CJ, Dejam A, Blood AB, Shields H, Kim-Shapiro DB, Machado RF, Tarekegn S, Mulla N, Hopper AO, Schechter AN, Power GG, Gladwin MT. Inhaled nebulized nitrite is a hypoxia-sensitive NO-dependent selective pulmonary vasodilator. Nat Med. 2004 Oct;10(10):1122-7. doi: 10.1038/nm1109. Epub 2004 Sep 12. PMID 15361865
- [Background] Kiowski W, Sutsch G, Hunziker P, Muller P, Kim J, Oechslin E, Schmitt R, Jones R, Bertel O. Evidence for endothelin-1-mediated vasoconstriction in severe chronic heart failure. Lancet. 1995 Sep 16;346(8977):732-6. doi: 10.1016/s0140-6736(95)91504-4. PMID 7658874
- [Background] Krowka MJ, Swanson KL, Frantz RP, McGoon MD, Wiesner RH. Portopulmonary hypertension: Results from a 10-year screening algorithm. Hepatology. 2006 Dec;44(6):1502-10. doi: 10.1002/hep.21431. PMID 17133488
- [Background] Lansley KE, Winyard PG, Bailey SJ, Vanhatalo A, Wilkerson DP, Blackwell JR, Gilchrist M, Benjamin N, Jones AM. Acute dietary nitrate supplementation improves cycling time trial performance. Med Sci Sports Exerc. 2011 Jun;43(6):1125-31. doi: 10.1249/MSS.0b013e31821597b4. PMID 21471821
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Effects of dietary nitrate on oxygen cost during exercise. Acta Physiol (Oxf). 2007 Sep;191(1):59-66. doi: 10.1111/j.1748-1716.2007.01713.x. Epub 2007 Jul 17. PMID 17635415
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Dietary nitrate reduces maximal oxygen consumption while maintaining work performance in maximal exercise. Free Radic Biol Med. 2010 Jan 15;48(2):342-7. doi: 10.1016/j.freeradbiomed.2009.11.006. Epub 2009 Nov 12. PMID 19913611
- [Background] Larsen FJ, Schiffer TA, Borniquel S, Sahlin K, Ekblom B, Lundberg JO, Weitzberg E. Dietary inorganic nitrate improves mitochondrial efficiency in humans. Cell Metab. 2011 Feb 2;13(2):149-59. doi: 10.1016/j.cmet.2011.01.004. PMID 21284982
- [Background] Mainguy V, Maltais F, Saey D, Gagnon P, Martel S, Simon M, Provencher S. Peripheral muscle dysfunction in idiopathic pulmonary arterial hypertension. Thorax. 2010 Feb;65(2):113-7. doi: 10.1136/thx.2009.117168. Epub 2009 Aug 30. PMID 19720606
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J; American College of Cardiology Foundation Task Force on Expert Consensus Documents; American Heart Association; American College of Chest Physicians; American Thoracic Society, Inc; Pulmonary Hypertension Association. ACCF/AHA 2009 expert consensus document on pulmonary hypertension a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association developed in collaboration with the American College of Chest Physicians; American Thoracic Society, Inc.; and the Pulmonary Hypertension Association. J Am Coll Cardiol. 2009 Apr 28;53(17):1573-619. doi: 10.1016/j.jacc.2009.01.004. No abstract available. PMID 19389575
- [Background] Mehta NJ, Khan IA, Mehta RN, Sepkowitz DA. HIV-Related pulmonary hypertension: analytic review of 131 cases. Chest. 2000 Oct;118(4):1133-41. doi: 10.1378/chest.118.4.1133. PMID 11035689
- [Background] Morrell NW, Adnot S, Archer SL, Dupuis J, Lloyd Jones P, MacLean MR, McMurtry IF, Stenmark KR, Thistlethwaite PA, Weissmann N, Yuan JX, Weir EK. Cellular and molecular basis of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S20-S31. doi: 10.1016/j.jacc.2009.04.018. PMID 19555855
- [Background] Mukerjee D, St George D, Coleiro B, Knight C, Denton CP, Davar J, Black CM, Coghlan JG. Prevalence and outcome in systemic sclerosis associated pulmonary arterial hypertension: application of a registry approach. Ann Rheum Dis. 2003 Nov;62(11):1088-93. doi: 10.1136/ard.62.11.1088. PMID 14583573
- [Background] Opravil M, Pechere M, Speich R, Joller-Jemelka HI, Jenni R, Russi EW, Hirschel B, Luthy R. HIV-associated primary pulmonary hypertension. A case control study. Swiss HIV Cohort Study. Am J Respir Crit Care Med. 1997 Mar;155(3):990-5. doi: 10.1164/ajrccm.155.3.9117037.
- [Background] Piazza G, Goldhaber SZ. Chronic thromboembolic pulmonary hypertension. N Engl J Med. 2011 Jan 27;364(4):351-60. doi: 10.1056/NEJMra0910203. No abstract available. PMID 21268727
- [Background] Ranque B, Authier FJ, Berezne A, Guillevin L, Mouthon L. Systemic sclerosis-associated myopathy. Ann N Y Acad Sci. 2007 Jun;1108:268-82. doi: 10.1196/annals.1422.029. PMID 17899625
- [Background] Rubin LJ; American College of Chest Physicians. Diagnosis and management of pulmonary arterial hypertension: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):7S-10S. doi: 10.1378/chest.126.1_suppl.7S. No abstract available. PMID 15249491
- [Background] Shorr AF, Helman DL, Davies DB, Nathan SD. Pulmonary hypertension in advanced sarcoidosis: epidemiology and clinical characteristics. Eur Respir J. 2005 May;25(5):783-8. doi: 10.1183/09031936.05.00083404. PMID 15863633
- [Background] Simonneau G, Robbins IM, Beghetti M, Channick RN, Delcroix M, Denton CP, Elliott CG, Gaine SP, Gladwin MT, Jing ZC, Krowka MJ, Langleben D, Nakanishi N, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S43-S54. doi: 10.1016/j.jacc.2009.04.012. PMID 19555858
- [Background] Sitbon O, Lascoux-Combe C, Delfraissy JF, Yeni PG, Raffi F, De Zuttere D, Gressin V, Clerson P, Sereni D, Simonneau G. Prevalence of HIV-related pulmonary arterial hypertension in the current antiretroviral therapy era. Am J Respir Crit Care Med. 2008 Jan 1;177(1):108-13. doi: 10.1164/rccm.200704-541OC. Epub 2007 Oct 11. PMID 17932378
- [Background] Smith AP, Demoncheaux EA, Higenbottam TW. Nitric oxide gas decreases endothelin-1 mRNA in cultured pulmonary artery endothelial cells. Nitric Oxide. 2002 Mar;6(2):153-9. doi: 10.1006/niox.2001.0400. PMID 11890739
- [Background] Souza R, Humbert M, Sztrymf B, Jais X, Yaici A, Le Pavec J, Parent F, Herve P, Soubrier F, Sitbon O, Simonneau G. Pulmonary arterial hypertension associated with fenfluramine exposure: report of 109 cases. Eur Respir J. 2008 Feb;31(2):343-8. doi: 10.1183/09031936.00104807. Epub 2007 Oct 24. PMID 17959632
- [Background] Tsihlis ND, Oustwani CS, Vavra AK, Jiang Q, Keefer LK, Kibbe MR. Nitric oxide inhibits vascular smooth muscle cell proliferation and neointimal hyperplasia by increasing the ubiquitination and degradation of UbcH10. Cell Biochem Biophys. 2011 Jun;60(1-2):89-97. doi: 10.1007/s12013-011-9179-3. PMID 21448667
- [Background] Uhlmann D, Ludwig S, Escher E, Armann B, Gabel G, Teupser D, Tannapfel A, Hauss J, Witzigmann H. Protective effect of a selective endothelin a receptor antagonist (BSF 208075) on graft pancreatitis in pig pancreas transplantation. Transplant Proc. 2001 Nov-Dec;33(7-8):3732-4. doi: 10.1016/s0041-1345(01)02523-4. No abstract available. PMID 11750590
- [Background] Weber C, Schmitt R, Birnboeck H, Hopfgartner G, van Marle SP, Peeters PA, Jonkman JH, Jones CR. Pharmacokinetics and pharmacodynamics of the endothelin-receptor antagonist bosentan in healthy human subjects. Clin Pharmacol Ther. 1996 Aug;60(2):124-37. doi: 10.1016/S0009-9236(96)90127-7. PMID 8823230
- [Background] Weitzenblum E, Chaouat A. Severe pulmonary hypertension in COPD: is it a distinct disease? Chest. 2005 May;127(5):1480-2. doi: 10.1378/chest.127.5.1480. No abstract available. PMID 15888814
- [Background] Hassoun, PM. Pulmonary arterial hypertension complicating connective tissue disease. In: Humbert M., Lynch JP, Eds. Pulmonary Hypertension. New York: Informa Healthcare USA, Inc. 2010: 161-175.
- [Background] Levi, DS, Scott, V, Aboulhosn J. Pulmonary arterial hypertension in congenital heart disease. In: Humbert, M, Lynch, JP, Eds. Pulmonary Hypertension. New York: Informa Healthcare USA, Inc. 2010: 176-195.
- [Background] Rubin LJ. Primary pulmonary hypertension. N Engl J Med. 1997 Jan 9;336(2):111-7. doi: 10.1056/NEJM199701093360207. No abstract available. PMID 8988890
- [Background] Shiva S. Mitochondria as metabolizers and targets of nitrite. Nitric Oxide. 2010 Feb 15;22(2):64-74. doi: 10.1016/j.niox.2009.09.002. Epub 2009 Sep 27. PMID 19788924
- [Background] Ware, JE et al. How to Score Version Two of the SF-36 Health Survey. Lincoln, RI: QualityMetric, Incorporated, 2000.